CLINICAL TRIAL: NCT03909984
Title: Promoting Implementation of Seizure Detection Devices in Epilepsy Care: the PROMISE Study
Brief Title: Promoting Implementation of Seizure Detection Devices in Epilepsy Care
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Epilepsie Instellingen Nederland (Other)
Collaborators: Kempenhaeghe Academic Center for Epileptology and Residential Epilepsy Care (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL62995.041.17
Record Dates: First submitted 2018-03-08; First posted 2019-04-10 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy in Children

STUDY DESIGN:
Intervention Model Description: Phase 1: Usual care (2 months), Phase 2: Intervention with monitoring true different devices (2 months), Phase 3: Optional phase with continued use of Nightwatch or tailoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): All participants will be monitored for 2 months.
  Interventions: Device: Nightwatch

INTERVENTIONS:
Device: Nightwatch — Nocturnal monitoring for 2 months with three different seizure detection devices.
  Other Names: Video and audio detection

SUMMARY:
This is a multicenter home-based medical device intervention study, with prospective validation of the wearable seizure detection device (Nightwatch) and retrospective validation of remote sensors (video and audio detection) in children. The investigators will also perform a feasibility and utility analysis of Nightwatch.

DETAILED DESCRIPTION:
Various remote and wearable sensor devices have become available for the detection of potentially dangerous seizures, with limited impact on epilepsy care so far. Both the investigator's remote and wearable seizure detection devices (SDDs) have been extensively tested and proven highly sensitive. Yet the home performance in children, an important target population, had been insufficiently studied.

Objective: 1. To test the performance of the wearable SDD (Nightwatch) prospectively and the remote SDD (automated video and audio analysis) retrospectively in children in a family home setting. 2. To assess the feasibility, cost-effectiveness and cost-utility of Nightwatch in children.

Study design: A multicenter home-based medical device intervention study with prospective validation of our wearable SDD.

Study population: 60 children (ages 4-16 years) with refractory epilepsy (≥1 major nocturnal seizure per week) recruited from the outpatient clinics of one of the participating epilepsy centers (Stichting Epilepsie instellingen Nederland (SEIN), Academic Centre of Epileptology Kempenhaeghe (Kempenhaeghe), University Medical Center Utrecht (UMCU)).

Intervention: Phase I: Two months of baseline (usual care); Phase 2: Two months of nocturnal seizure monitoring at home, using Nightwatch and the remote SDD.

Main study parameters/endpoints: The diagnostic performance of Nightwatch and the remote SDD algorithms, i.e. sensitivity, positive predictive value, false alarm rate and % time with uninterrupted signal output. The investigators will evaluate feasibility of Nightwatch through surveys on quality of life, sleep, parental strain, interviews with parents/guardians and neurologists, and a value sensitive design group session. The investigators will also perform a cost-effectiveness and cost-utility analysis by medical consumption and costs questionnaires.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Implementing SDDs will not pose any direct or substantial risk. Study participation can be a burden though, due to impact of the devices on privacy, number of false alarms and time spent on the questionnaires and interviews. Application of the SDDs, however, might offer better insight into the actual number of nocturnal seizures in a child, change in medical management and facilitate appropriate interventions in major motor seizures. If reliable, SDDs may improve the night rest of both patient and parents/guardians.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-16 years
* Diagnosis of refractory epilepsy with ≥1 major nocturnal seizure per week.
* Treated at one of the following epilepsy centers: SEIN, Kempenhaeghe or UMCU.
* Written informed consent by legal representatives (mostly parents) and also by the subject when aged ≥12 years and capable of signing informed consent.

Exclusion Criteria:

* Intensive non-epileptic movement patterns such as severe choreatiform movements, intensive sleep walking, or frequent night terrors (> 1/week).
* Minor motor seizures only, i.e. non-generalized or short (< 10 sec.) tonic seizures or isolated myoclonias that are self-limited and do not require intervention.
* Presence of a pacemaker or cardiac arrhythmias that may generate false alarms (e.g. supraventricular tachycardia).
* Inability to comply to the trial procedure.
* Skin characteristics (e.g. tattoo) that may affect photoplethysmography and thereby influence performance of the Nightwatch.
* Dependence on another SDD (e.g. Emfit or saturation monitor). Simultaneous use of a baby phone (or other types of microphones) is permitted.
* Subjects who are not sleeping alone in the bed (i.e. co-sleeping in the parents'/guardians' bed influences the remote SDD). Subjects and parents/guardians are not allowed to change their sleeping habits for the duration of the study only.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance Nightwatch - sensitivity | Monitoring period of 2 months per participant.
  Performance of Nightwatch to detect major nocturnal motor seizures in children at home, measured prospectively by means of sensitivity.
Diagnostic performance Nightwatch - positive predictive value | Monitoring period of 2 months per participant.
  Performance of Nightwatch to detect major nocturnal motor seizures in children at home, measured prospectively by means of positive predictive value.
Diagnostic performance Nightwatch - false alarm rate | Monitoring period of 2 months per participant.
  Performance of Nightwatch to detect major nocturnal motor seizures in children at home, measured prospectively by means of false alarm rate.
Diagnostic performance Nightwatch - % time with uninterrupted signal | Monitoring period of 2 months per participant.
  Performance of Nightwatch to detect major nocturnal motor seizures in children at home, measured prospectively by means of % of time with uninterrupted signal output.

SECONDARY OUTCOMES:
Diagnostic performance of video and audio detection - sensitivity | Monitoring period of 2 months per participant.
  Diagnostic performance of our remote seizure detection devices (video and audio) to detect major nocturnal motor seizures in children at home, measured retrospectively by means of sensitivity.
Diagnostic performance of video and audio detection - positive predictive value | Monitoring period of 2 months per participant.
  Diagnostic performance of our remote seizure detection devices (video, audio) to detect major nocturnal motor seizures in children at home, measured retrospectively by means of positive predictive value.
Diagnostic performance of video and audio detection - false alarm rate | Monitoring period of 2 months per participant.
  Diagnostic performance of our remote seizure detection devices (video, audio) to detect major nocturnal motor seizures in children at home, measured retrospectively by means of false alarm rate.
Diagnostic performance of video and audio detection - % time with uninterrupted signal output. | Monitoring period of 2 months per participant.
  Diagnostic performance of our remote seizure detection devices (video, audio) to detect major nocturnal motor seizures in children at home, measured retrospectively by means of % time with uninterrupted signal output.
Feasibility of Nightwatch will be examined in an interview with parents/guardians, focussing on different aspects of the device. | 4 month period (2 months usual care + 2 months monitoring)
  Feasibility of Nightwatch with a mixed methods approach focusing on Acceptability, Demand, Implementation, Practicality, Expansion, Limited-efficacy testing, impact of the SDD on parents/guardians with children (interview).
Feasibility of Nightwatch by means of Caregiver Strain Index (CSI). | 4 month period (2 months usual care + 2 months monitoring)
  Effect of Nightwatch on parental stress, with a stress questionnaire (CSI), containing 13 questions about stress with 'yes/no' answers.
  11-13 tims 'yes' indicates high level of stress, 7-10 times 'yes' indicates medium level of stress and 0-6 times 'yes' means low level of stress.
Feasibility of Nightwatch by means of Pittsburgh Sleep Quality Index (PSQI). | 4 month period (2 months usual care + 2 months monitoring)
  Effect of Nightwatch on parental sleep with a sleep questionnaire (PSQI), containing 10 questions about sleep, with scales from 1-4 to indicate how often parents/guardians experience certain sleep problems.
Feasibility of Nightwatch by means of the Quality of Life questionnaire: EQ-5D-5L | 4 month period (2 months usual care + 2 months monitoring)
  Effect of Nightwatch on parental quality of life, with a QoL questionnaire (EQ-5D-5L), containing 5 questions about the person's health with a 1-5 scale indicating the severity of a certain health problem and a 0-100 rating scale of their health.
Cost-effectiveness analysis of Nightwatch | 4 month period (2 months usual care + 2 months monitoring)
  Economic evaluation from a societal prospective of Nightwatch involving a cost-effectiveness analysis (CEA).
Cost-utility analysis of Nightwatch | 4 month period (2 months usual care + 2 months monitoring)
  Economic evaluation from a societal prospective of Nightwatch involving a cost- a cost-utility analysis (CUA).

CONTACTS AND LOCATIONS:
Overall Officials: Anouk van Westrhenen, MD, Principal Investigator — Stichting Epilepsie Instellingen Nederland; Roland D Thijs, MD, PhD, Study Director — Stichting Epilepsie Instellingen Nederland
Locations (3):
- Netherlands (3):
  - Stichting Epilepsie Instellingen Nederland (SEIN), Heemstede, Achterweg 5
  - Academic Center of Epileptology Kempenhaeghe, Heeze
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Principal investigators will share necessary information on participants and enrollment.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] van Westrhenen A, Lazeron RHC, van Dijk JP, Leijten FSS, Thijs RD; Dutch TeleEpilepsy Consortium. Multimodal nocturnal seizure detection in children with epilepsy: A prospective, multicenter, long-term, in-home trial. Epilepsia. 2023 Aug;64(8):2137-2152. doi: 10.1111/epi.17654. Epub 2023 Jun 14. PMID 37195144

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03909984/Prot_SAP_000.pdf